CLINICAL TRIAL: NCT05280366
Title: A Prospective, Randomized, Multi-center Evaluation of the Safety and Effectiveness of the STREAMLINE®SURGICAL SYSTEM Compared to iStent Inject W® in Patients With Open-Angle Glaucoma
Brief Title: STREAMLINE®SURGICAL SYSTEM Compared to iStent Inject W® in Patients With Open-Angle Glaucoma
Acronym: VENICE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New World Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF6-CL-21-02
Record Dates: First submitted 2021-12-29; First posted 2022-03-15 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-04

CONDITIONS: Open Angle Glaucoma
Keywords: glaucoma; Goniotomy; MIGS
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Streamline Surgical System (Other): Streamline Surgical System procedure administered
  Interventions: Device: Streamline Surgical System
- iStent Inject W (Active Comparator): iStent Inject W implanted
  Interventions: Device: iStent Inject W

INTERVENTIONS:
Device: Streamline Surgical System — Completion of the Streamline Surgical System procedure
  Arms: Streamline Surgical System
Device: iStent Inject W — Implantation of competitor device
  Arms: iStent Inject W

SUMMARY:
A study of the Streamline Surgical System versus competitor

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of Mild to Moderate Primary Open Angle Glaucomma

Exclusion Criteria:

* Other types of glaucoma including but not limited to: Normal tension glaucoma, pseudoexfoliative glaucoma, narrow angle glaucoma, traumatic, congenital, malignant, uveitic or neovascular glaucoma. Ocular hypertension.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in mean unmedicated diurnal Intraocular Pressure (IOP) | 24 months
  Change in mean unmedicated diurnal Intraocular Pressure (IOP) over time

CONTACTS AND LOCATIONS:
Overall Officials: Elysia Ison, OD, Study Director — New World Medical, Inc.
Locations (20):
- United States (18):
  - Vold Vision, Fayetteville, Arkansas
  - Visionary Research Institute, Newport Beach, California
  - Wolstan and Goldberg Eye Associates, Torrance, California
  - University of Colorado, Aurora, Colorado
  - Ocala Eye, Ocala, Florida
  - Georgia Eye Partners, Atlanta, Georgia
  - The Eye Institute, Louisville, Kentucky
  - Ophthalmology Associates, St Louis, Missouri
  - Eye Associates of North New Jersey, Dover, New Jersey
  - Eye Associates Surgical Center, Vineland, New Jersey
  - Ross Eye Institute, Orchard Park, New York
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - University Eye Specialists, Maryville, Tennessee
  - Ophthalmology Associates, Fort Worth, Texas
  - Berkely Eye Center, Houston, Texas
  - R & R Eye Research, San Antonio, Texas
  - Piedmont Eye Center, Lynchburg, Virginia
  - Eye Centers of Racine and Kenosha, Racine, Wisconsin
- Clinica 20/20, San José, Costa Rica
- Clinica Laser y Ultrasonido Ocular, Puebla City, Mexico

IPD SHARING:
Plan to Share IPD: No